CLINICAL TRIAL: NCT03513887
Title: Noninvasive Tests to Predict the Presence of Esophageal Varices in Patients With Liver Cirrhosis
Status: Completed | Type: Observational
Sponsor: Second Affiliated Hospital of Xi'an Jiaotong University (Other)
Responsible Party: Sponsor
Other Study IDs: 2018016
Record Dates: First submitted 2018-03-29; First posted 2018-05-02 (Actual); Last update posted 2019-05-29 (Actual); Status verified 2018-02

CONDITIONS: Cirrhosis
Keywords: cirrhosis,varices,variceal bleeding, noninvasive tests,TE
MeSH Terms: conditions — Fibrosis

STUDY DESIGN:
Observational Model: Case-Crossover | Time Perspective: Cross-Sectional
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (1):
- Group/Cohorts: we will prospectively collect patients with liver cirrhosis who fulfill all inclusion criterias and will be treated in the Department of Gastroenterology of the Second Affiliated Hospital of Xi'an Jiaotong University.

SUMMARY:
Liver cirrhosis is caused by chronic liver diseases, varices exist in 30 - 60% of patients with liver cirrhosis. Variceal bleeding is one of the most important complications of cirrhosis, accelerating the progression of decompensation to a stage at which the patient is at an extremely high risk of death. Endoscopy is the gold standard for the diagnosis of varices, However, periodic endoscopic screening in all cirrhotic patients might unnecessarily induce an invasive and expensive procedure, ultimately increasing not only the medical workload of endoscopy units, but also the financial burden of patients. To avoid unnecessary endoscopy in low- risk patients, some simple, non-invasive and accurate tests have been developed to identify EVs. Such as Transient elastography (TE) , which is a noninvasive tool that measures liver stiffness (LS) correlating to liver fibrosis stage. Moreover, the LS-spleen size-to-platelet ratio score (LSPS), which is a combination of three simple examination methods (LS, spleen size and platelet count) has been established to accurately predict EVs in patients with cirrhosis. Therefore, investigators design this cross-sectional study to assess these non-invasive tests in predicting the presence of EVs in patients with cirrhosis.

DETAILED DESCRIPTION:
Liver cirrhosis is a result of excessive extracellular matrix deposition in the liver in response to chronic inflammatory injury triggered by chronic liver diseases. And Cirrhosis is classified in 2 distinct clinical stages, compensated (Currently, both terms : "compensated advanced chronic liver disease(cACLD)" and "compensated cirrhosis" are acceptable) and decompensated, defined by the presence or absence of overt clinical complications of cirrhosis (ascites, variceal hemorrhage, hepatic encephalopathy). Portal hypertension is a frequent complication of liver cirrhosis, a contributing fator for ascites and hepatic encephalopathy, and a direct cause of variceal hemorrhage. An increase in portal pressure leads to the development of portosystemic collateral circulation, of which varices are the most important clinical feature. In accordance with the Baveno II consensus conference, esophageal varices (EVs) were classified as absent, small (diameter < 5 mm) or large (diameter ≥ 5 mm). The presence of red wale marks on the variceal wall in EVs was also recorded. EVs at a high risk for bleeding were defined according to the Baveno V criteria as large EVs or small EVs with red signs or EVs in patients with Child-Pugh class C disease. varices exist in 30 - 60% of patients with liver cirrhosis, depending on the severity of Portal hypertension. The yearly rate of development of new cases is 5 - 10% , whereas the growth rate from small to large varices ranges between 5 and 30 %.

Variceal bleeding is the most important and the most lethal complication of cirrhosis, accelerating the progression of decompensation to a stage at which the patient is at an extremely high risk of death. Therefore, the diagnosis, prevention, and management of EVs are important for patients with cirrhosis. And screening for EVs in all patients with cirrhosis is also strongly recommended across guidelines and consensus statements. Endoscopy is the gold standard for the diagnosis of varices, and is recommended as the screening method to identify those who should undergo prophylactic treatment when the diagnosis of cirrhosis is made. Nonselective β-blockers significantly reduce the bleeding rate in more than half of patients with high-risk EVs (HEVs). However, as the prevalence of HEVs at any given point in time is 15 - 25%, the majority of subjects undergoing screening endoscopy either do not have varices, or have varices that do not require prophylactic therapy. Therefore, periodic endoscopic screening in all cirrhotic patients, especially low-risk groups, might unnecessarily induce an invasive and expensive procedure, ultimately increasing not only the medical workload of endoscopy units, but also the financial burden to patients, as the number of patients with chronic liver disease increases and their survival improves. Furthermore, compliance may be limited, because even asymptomatic patients may be required to repeatedly undergo an unpleasant endoscopic procedure, which usually requires conscious sedation decreasing work productivity, It also carries rare but serious complications. Patients might be reluctant to receive endoscopy and become discouraged in starting preventive measures. All of these reasons lead to decline in patient compliance with treatment and follow-ups. Meanwhile, the endoscopy-related complications reported by a related article is close to 0.1% of incidence.

To avoid unnecessary endoscopy in low-risk patients, some simple, non-invasive and accurate tests have been developed to identify EVs. Transient elastography (TE) is a noninvasive tool that measures liver stiffness (LS) correlating to liver fibrosis stage. While LS also shows potential in the prediction of EVs, its role is still under debate. Moreover, the LS-spleen size-to-platelet ratio score (LSPS), which is a combination of three simple examination methods (LS, spleen size and platelet count) has been established to accurately predict EVs in patients with cirrhosis. And recent Baveno VI recommended the combination of transient elastography and platelet count for ruling out HEVs in patients with chronic liver disease.

Although there is a correlation between these non-invasive tools and the presence of EVS or HEVs, the optimal cut-offs and their validities vary in the different studies with different etiologies. In addition, the qualities of EVs assessment have not been provided in these studies. Therefore, investigators design this cross-sectional study to assess these non-invasive tests in predicting the presence of EVs in patients with cirrhosis. This could prevent unnecessary endoscopy with related complications and costs. And the results of noninvasive tests will be compared with endoscopy (ie, the gold standard for diagnosing EVs).

ELIGIBILITY:
Inclusion Criteria:

1. Aged 18 - 80 years old;
2. Diagnosis of liver cirrhosis (Cirrhosis is diagnosed using standard laboratory, radiological, and physical examination findings, or by liver histology in equivocal cases);
3. Paired noninvasive tests (blood tests, TE, abdominal CT, and/or ultrasound) and endoscopy within 3 months;

Exclusion Criteria:

1. A body mass index > 35;
2. Severe cardiopulmonary diseases, renal failure，acute illness; infectious diseases;
3. Pregnant or breast-feeding subjects;
4. Previous splenectomy or liver transplantation;(文献55)
5. Previous β-blocker therapy;
6. Endoscopic treatments (band ligation or sclerotherapy);
7. Previous surgery for portal hypertension or transjugular intrahepatic portosystemic stent shunt placement;
8. Portal vein or splenic vein thrombosis;
9. Current or past history of hepatocellular carcinoma;
10. Presence of severe ascites that might significantly hamper the accurate assessment of LSM;
11. Unreliable LSM with an interquartile range (IQR) to median value ratio (IQR/M) of > 0.3, a success rate of < 60% , or validated measurements of < 10;

Ages: 18 Years to 80 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: In this cross-sectional study, we will prospectively collect patients with liver cirrhosis who fulfill all inclusion criterias and will be treated in the Department of Gastroenterology of the Second Affiliated Hospital of Xi'an Jiaotong University from March 2018 to December 2018.
Sampling Method: Non-Probability Sample
Enrollment: 111 (Actual)
Dates: Start 2018-02-28 (Actual); Primary Completion 2019-01-12 (Actual); Study Completion 2019-01-12 (Actual)

PRIMARY OUTCOMES:
EVs and HEVs detected by endoscopy | 3 months
  All patients will undergo or have been undergone endoscopy, endoscopy is performed by a small number of experienced endoscopy operators. The severity of varices and the presence of red signs will be recorded.

CONTACTS AND LOCATIONS:
Overall Officials: Jinhai Wang, Study Director — The Second Affiliated Hospital of Xi'an Jiaotong University,Xi'an, Shaanxi, China
Locations (1):
- The second affiliated hospital of xi'an jiaotong university, Xi'an, Shaanxi, China